CLINICAL TRIAL: NCT03473678
Title: Influence of Dietary Nitrate Supplementation on Blood Pressure, Walking Economy, Functional Physical Capacity and Cognitive Function in Healthy Older Adults
Brief Title: Dietary Nitrate and Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 121964
Record Dates: First submitted 2018-01-31; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Blood Pressure; Cognitive Change; Functional Capacity; Brain Metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): 2 x 70mL concentrated juice per day for 10 days
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): 2 x 70mL concentrated juice per day for 10 days
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — concentrated beetroot juice
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — concentrated beetroot juice
  Arms: Nitrate-depleted beetroot juice

SUMMARY:
This study investigates the influence of dietary nitrate supplementation on cardiovascular health and physical and cognitive performance in older adults. Participants will receive both a nitrate containing beetroot juice for 10 days and a nitrate depleted beetroot juice for 10 days

DETAILED DESCRIPTION:
A recent exciting finding is that dietary nitrate supplementation (in the form of beetroot juice) appears to reduce the amount of oxygen needed to complete moderate intensity walking in healthy, young individuals. Nitrate is known to be converted in the body to nitric oxide (NO), a substance which reduces blood pressure and may affect the energy-producing mechanisms inside muscle cells. Exercise tolerance and muscle function typically declines with age and nitrate supplementation therefore may help improve cardiovascular health and the ability to carry out low-intensity daily activities in aging populations. The purpose of this study is to see if healthy, elderly individuals benefit from beetroot juice intake similarly to the effects seen in young adults. If this is indeed the case, then it may suggest that dietary supplementation with a relatively cheap, widely available, and natural food product may improve the ability of healthy elderly individuals to undergo everyday tasks and ultimately improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 70 - 80 years of age
2. male or female

Exclusion Criteria:

1. involved in regular structured exercise
2. receiving medication for:

   * pulmonary conditions
   * cardiovascular conditions
   * metabolic conditions
   * musculoskeletal conditions
   * ulcerative colitis
   * renal disease

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-12 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 10 days
  Change in blood pressure between interventions

SECONDARY OUTCOMES:
Oxygen cost of exercise | 10 days
  Change in oxygen consumption during exercise
Serial Subtraction test | 10 days
  change in performance of the Serial Subtraction test
Microbiome | 10 days
  change in oral microbiome measured by sequencing bacterial 16S rRNA genes
Brain metabolism | 10 days
  change in brain metabolites measured measured by 1H MRS
6 minute walk test | 10 days
  change in performance of 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Jones, PhD, Principal Investigator — University of Exeter
Locations (1):
- Sport and Health Sciences, University of Exeter, Exeter, Devon, United Kingdom